CLINICAL TRIAL: NCT00379431
Title: A Protocol Based Treatment for Early and Severe Systemic Sclerosis With (Anti-CD20), Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/257
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Early and Severe Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administration of rituximab and methylprednisolone (Experimental)
  Interventions: Drug: Administration of rituximab and methylprednisolone

INTERVENTIONS:
Drug: Administration of rituximab and methylprednisolone — Rituximab:
  Pharmaceutical form: Concentrate for solution for infusion. Maximum duration of treatment: 28 weeks Maximum dose allowed: 2000 mg (use of total dose) Route of administration: intravenous use.

SUMMARY:
Rituximab 1000 mg i.v. will be given on day 1 and 15, week 26 - 28, together with a corticosteroid regimen consisting of methylprednisolone 100 mg i.v. 30 minutes prior to both infusions.

ELIGIBILITY:
Inclusion Criteria:

* male or female >= 18 years
* SSc according to the ARA criteria for systemic sclerosis
* Disease duration less than 4 years (from the appearance of skin changes (oedema, fibrosis)
* Inadequate response to methotrexate (at least 12 weeks 10 mg/w, except if not tolerated
* Antibodies specific for systemic sclerosis: anti-topoisomerase; anti-centromere antibodies
* Severe disease defined by either one of the following: a modified Rodnan skin score (TSS° >= 14 ), disease activity score >= 3
* Contraception for women with childbearing potential. Sexual abstinence is an alternative to contraception.
* Patient has signed informed consent.

Exclusion Criteria:

* disease duration more than 4 years
* FVC <= 50%
* LVEF <= 40% of predicted value
* DLCO <= 40% of predicted value
* Lack of peripheral venous access
* Pregnancy or breast feeding
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease), evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine or gastrointestinal disorders which, in the investigator's opinion, would preclude patient participation
* Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection.
* Known active infection of any kind (excluding fungal infections of mail beds), or any major episode of infection requiring hospitalization or treatment with i.v. anti-infectives within 4 weeks of baseline or completion of oral anti-infectives within 2 weeks prior to baseline.
* History of deep space/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks prior to baseline.
* History of serious recurrent or chronic infection (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks prior to screening).
* History of cancer, including solid tumors, hematologic malignancies and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured).
* History of a severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of rituximab or to murine proteins.
* Concurrent treatment with any biologic agent or DMARD other than MTX. Treatment must be discontinued 14 days prior to baseline , except for the following: azathioprine for ≥ 28 days; leflunomide for ≥ 8 weeks (or ≥ 14 days after 11 days of standard cholestyramine or activated charcoal washout); infliximab ≥ 8 weeks; adalimumab ≥ weeks.
* Previous treatment with > 1 biological agent.
* Previous treatment with any cell depleting therapies, including investigational agents.
* Treatment with any investigational agent within 28 days of baseline or 5 half-lives of the investigational drug (xhich ever is the longer).
* Receipt of any vaccine within 28 days prior to baseline
* Intolerance or contraindications to i.v. glucocorticoids.
* Positive serum human chorionic gonadotropin (hCG) measured at screening or a positive pregnancy test prior to the first rituximab infusion.
* Positive tests for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C serology.
* Hemoglobin < 8.0 g/dL.
* Concentrations of serum IgG and/or IgM below 5.0 and 0.40 mg/mL, respectively.
* Absolute neutrophil count (ANC) < 1.5 X 10³/µL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-11-27 (Actual); Primary Completion 2009-02-02 (Actual); Study Completion 2009-02-02 (Actual)

PRIMARY OUTCOMES:
Death | 28 weeks
Heart failure defined as a LVEF< 30% | 28 weeks
Lung failure defined as a resting PaO2< 60mmHg | 28 weeks
Evolution of antibody titers. | 28 weeks
Deterioration, improvement or stabilisation of, disease activity score, 6-m walking distance, SHAQ, LVEF and creatinine clearance | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Filip De Keyser, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - UCL St. Luc Brussel, Brussels
  - UZ Brussel, Brussels
  - University Hospital Ghent, Ghent
  - UZ Gasthuisberg Leuven, Leuven

REFERENCES:
- [Derived] Melsens K, De Keyser F, Decuman S, Brusselle G, De Pauw M, Deschepper E, De Wilde K, Elewaut D, Piette Y, Vandecasteele E, Smith V. Assessment of sensitivity to change of the European Scleroderma Study Group activity index. Clin Exp Rheumatol. 2016 Sep-Oct;34 Suppl 100(5):148-151. Epub 2016 Jul 18. PMID 27463733
- [Derived] Smith V, Pizzorni C, Riccieri V, Decuman S, Brusselle G, DE Pauw M, Deschepper E, Piette Y, Ruaro B, Sulli A, Vandecasteele E, Melsens K, DE Keyser F, Cutolo M. Stabilization of Microcirculation in Patients with Early Systemic Sclerosis with Diffuse Skin Involvement following Rituximab Treatment: An Open-label Study. J Rheumatol. 2016 May;43(5):995-6. doi: 10.3899/jrheum.151018. No abstract available. PMID 27134280
- [Derived] Bonroy C, Smith V, Deschepper E, De Keyser F, Devreese K. Specific Antinuclear Antibody Level Changes after B Cell Depletion Therapy in Systemic Sclerosis Are Associated with Improvement of Skin Thickening. J Rheumatol. 2016 Jan;43(1):247-9. doi: 10.3899/jrheum.150105. No abstract available. PMID 26724322
- [Derived] Smith V, Piette Y, van Praet JT, Decuman S, Deschepper E, Elewaut D, De Keyser F. Two-year results of an open pilot study of a 2-treatment course with rituximab in patients with early systemic sclerosis with diffuse skin involvement. J Rheumatol. 2013 Jan;40(1):52-7. doi: 10.3899/jrheum.120778. Epub 2012 Nov 1. PMID 23118116
- [Derived] Smith V, Van Praet JT, Vandooren B, Van der Cruyssen B, Naeyaert JM, Decuman S, Elewaut D, De Keyser F. Rituximab in diffuse cutaneous systemic sclerosis: an open-label clinical and histopathological study. Ann Rheum Dis. 2010 Jan;69(1):193-7. doi: 10.1136/ard.2008.095463. PMID 19103636
- See also: Website University Hospital Ghent — http://www.uzgent.be